CLINICAL TRIAL: NCT05123677
Title: Serial Maternal Haemodynamic Monitoring in Pregnancy for the Prediction of Pre-eclampsia and Fetal Growth Restriction in a High-risk Population
Brief Title: Cardiac Output Monitoring to Predict Pre-Eclampsia and Restricted Growth (COMPaRE)
Acronym: COMPaRE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Nadiah Hashim Arrifin, Fetal Medicine Clinical Research Fellow, Sandwell & West Birmingham Hospitals NHS Trust
Other Study IDs: 21MATE01
Record Dates: First submitted 2021-10-28; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Fetal Growth Retardation; Pre-Eclampsia
MeSH Terms: conditions — Fetal Growth Retardation; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Risk: These patients are screened to be low-risk for pre-eclampsia and fetal growth restriction by the guidelines set out by the National Institute for Health and Care Excellence; and the Royal College of Obstetricians & Gynaecologists, respectively.
  Interventions: Diagnostic Test: Non-invasive haemodynamic assessment; Diagnostic Test: Maternal ophthalmic artery doppler
- High Risk: These patients are screened to be high-risk for pre-eclampsia and fetal growth restriction by the guidelines set out by the National Institute for Health and Care Excellence; and the Royal College of Obstetricians & Gynaecologists, respectively.
  Interventions: Diagnostic Test: Non-invasive haemodynamic assessment; Diagnostic Test: Maternal ophthalmic artery doppler

INTERVENTIONS:
Diagnostic Test: Non-invasive haemodynamic assessment — Maternal non-invasive haemodynamic assessment: a pressure cuff (similar to the one used to measure blood pressure) is applied to the arm and thigh, and a further neck sensor applied. Information about the function of heart and major blood vessels are recorded
Diagnostic Test: Maternal ophthalmic artery doppler — Maternal ophthalmic artery doppler: an ultrasound probe is applied gently over the eyelid for a few seconds to study the blood flow of the main artery to the eye

SUMMARY:
Pre-eclampsia (PET) and fetal growth restriction (FGR) are common complications of pregnancy that affect up to 15% of pregnancies in the UK. These conditions can have potentially devastating consequences to mothers and babies in pregnancy. Pre-term birth, that is often medically indicated to treat severe PET and FGR can cause cerebral palsy, breathing difficulty, developmental delay and even death in affected babies. Mothers who suffer from PET are at risk of seizures, strokes, multi-organ failure and future chronic hypertension. It is now thought that PET and FGR may result from poor adaptation of the maternal cardiovascular system to normal pregnancy. This project aims to study the patterns within the maternal cardiovascular system and haemodynamic profile in women who are at high risk of PET and FGR by using non-invasive methods to gather information about the functions of their hearts and major blood vessels. The investigators hope to elucidate the patterns that may offer an early warning to mothers who may develop PET and whose fetuses may be growth restricted. This would be an opportunity to more closely monitor, modify risk factors and treat earlier women who develop these conditions. Women who are at a high risk of PET and FGR as stipulated in the relevant Royal College of Obstetrics & Gynaecology and National Institute of Clinical Excellence guidelines and who give their consent will be eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged ≥18 at time of conception
* Case subjects are at high risk of PET by NICE guidelines ( ≥1 high risk factor or >1 moderate risk factor) or high risk of SGA by RCOG Guidelines (≥1 major risk factor or ≥3 minor risk factors). Control subjects do not meet this criteria

Exclusion Criteria:

* Maternal age <18 years of age at time of booking
* Fetal structural or genetic abnormality
* Multiple pregnancy
* Known underlying maternal cardiac condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant patients who book in the first trimester at Birmingham City Hospital within the specified study dates.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of pre-eclampsia | From 20 weeks gestation to 12 weeks post-partum.
  This is defined as hypertension of >140/90 mmHg and significant proteinuria. This is defined as urinalysis showing proteinuria of >1+ or laboratory-quantified urine protein:creatinine ratio of >30mg/mmol. These are assessed at every study visit.
Diagnosis of fetal growth restriction | From 20 weeks gestation to birth.
  This is diagnosed on ultrasound or at birth. During ultrasound scans at visits 2 and 3, fetal weight is estimated using the Hadlock formula from measurements of the fetal abdominal circumference, femur length and head circumference. This is then plotted onto customised growth chart. Fetal growth restriction is diagnosed antenatally when the estimated fetal weight is under the 3rd centile or under the 10th centile in the presence of abnormal ultrasound dopplers. Abnormal ultrasound dopplers are defined as raised pulsatility index in the fetal umbilical artery, middle cerebral artery or ductus venosus. At birth, fetal growth restriction is diagnosed when the measured birthweight plots under the 10th centile on the customised growth chart.

SECONDARY OUTCOMES:
Pregnancy outcome | From birth to 12 weeks of age
  This is concerned with the 3 possible outcomes of the pregnancy: livebirth, stillbirth or neonatal death.
Gestational age at delivery | At delivery
  This is the recorded age of gestation at the time of delivery, in weeks and days
Birthweight centile | At birth
  This is a measure of the baby's weight at birth, in grams. This is then plotted onto a customised growth chart, accounting for maternal ethnicity and body mass index.
Duration of neonatal unit admission | At delivery
  This is concerned with whether the baby is admitted to the neonatal admission unit following delivery. If admitted, duration would be quantified in days and hours.
Intrapartum or immediate postpartum complications. | From the onset of active labour (4cm cervical dilatation and regular contractions of 3-4:10 minutes) till 48 hours post-delivery
  This is concerned with the development of complications in the mother, in relation to haemorrhage and hypertensive disorders.
Persistence of maternal haemodynamic changes | 6-12 weeks postpartum (during study visit 4)
  Maternal haemodynamic changes assessed postpartum showing the persistence of haemodynamic changes noted antenatally

IPD SHARING:
Plan to Share IPD: No